CLINICAL TRIAL: NCT05413187
Title: A Double-Blind, Placebo Controlled, Randomized Trial to Assess the Efficacy and Safety of Medical Grade Cannabis (MGC) in Children Diagnosed With Autism Spectrum Disorder
Brief Title: A Trial to Assess the Efficacy and Safety of Medical Grade Cannabis in Children Diagnosed With Autism Spectrum Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn due to COVID-19
Sponsor: TO Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SCRC17039
Record Dates: First submitted 2019-04-24; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Autistic Disorder
Keywords: Cannabis; Autism
MeSH Terms: conditions — Autistic Disorder; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Approximately forty children between the ages of two to eight years old with a documented diagnosis of Autism.
  The trial population will be randomized in a 1:1 ratio.
Who Masked: Participant, Investigator
Masking Description: During the trial procedures, SCRC coordinators and the sponsors will be exposed to the trial randomization. All other personnel including principle investigator, investigators, research assistants etc. will be blinded to the randomization and trial arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Grade Cannabis oil 30% CBD ,1.5% Δ9-THC (Active Comparator): during phase 1; subjects will receive cannabis oil. They will receive treatment for twelve weeks, following a four-week washout period without any treatment. In the second phase, a crossover of trial arms will take place and patients who received cannabis oil will then receive placebo and vice versa. Clinical evaluation will take place after completing each phase.
  Interventions: Drug: Medical Grade Cannabis oil
- Olive oil and Chlorophyl (Placebo Comparator): during phase 1; subjects will receive placebo. They will receive treatment for twelve weeks, following a four-week washout period without any treatment. In the second phase, a crossover of trial arms will take place and patients who received cannabis oil will then receive placebo and vice versa. Clinical evaluation will take place after completing each phase.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Medical Grade Cannabis oil — MGC, 30% CBD and 1.5% Δ9-THC
  Other Names: Cannabis oil
  Arms: Medical Grade Cannabis oil 30% CBD ,1.5% Δ9-THC
Drug: Placebos — Olive oil and Chlorophyl
  Arms: Olive oil and Chlorophyl

SUMMARY:
This single center, double-blinded, randomized, placebo-controlled crossover trial will assess the efficacy and safety of extraction of cannabis flowers dissolved in olive oil (30% CBD and 1.5% Δ9-THC) vs. placebo in patients diagnosed with Autism Spectrum Disorder. The trial will contain two phases in which patients will first receive a twelve-week treatment of either cannabis or placebo followed by four weeks wash out period and another twelve weeks of crossover in the trial arms.

DETAILED DESCRIPTION:
Visit 1 - Screening and Enrollment The screening and enrollment procedures will take place at the Preschool Psychiatric Unit in Soroka University Medical Center (SUMC). Parents of children who meet all inclusion criteria and none of the exclusion criteria will be offered to participate in this trial. Interested parents will sign an informed consent form (ICF) and receive a copy. A medical cannabis license request will be sent to the Medical Cannabis Unit ("Yakar") for cannabis treatment for the child and upon approval the patient will be enrolled to the trial.

Medical history will be assessed, patients who do not have a general and neurologic exam during the past year previous to the initiation of the trial will be referred to their physician. Clinical and behavioral assessment will be performed by the investigator, vital signs and weight and height will be measured, and a urine sample will be taken. All concomitant medication taken by the patient will be documented.

The YAKAR's medical cannabis license application form and a confidentiality waiver form will be sent to the YAKAR. The physician will explain to the patient the medical license conditions and that the patient's participation in the trial can be terminated at any time.

Visit 2 - Randomization and Initiation of Phase 1 When the medical cannabis license arrives, a copy of the patient's license will be included into the trial source documents. Prior to randomization inclusion and exclusion criteria will be re-assessed to make sure the patient is eligible to participate in the trial.

A clinical and behavioral evaluation will be held by the investigator and will also include the following questionnaires:

* The Aberrant Behavior Checklist-Community (ABC-C)
* The Children's Sleep Habit Questionnaire (CSHQ)
* Sensory Profile II (SP-2) Questionnaire A urine sample will be taken for the presence of cannabis. The patient will participate in a 10-minute eye tracking test. A detailed guidance and instructions on the use of the IP at home will be given by a member of the trial team.The IP (drug or placebo based upon randomization) will be administered to the parents. The first dose administration will take place in the morning after the visit.

A compliance diary will be handed out to the parents and they will be instructed to fill out the daily administration of the IP.

Visit 3 (week 6 ± 5 days) Mid Phase 1 During this visit, a clinical and behavioral evaluation will be held via questionnaires (ABC-C, CGI-1) and the investigator. The patient compliance diary will be reviewed and returned to the parents for further documentation. Adverse events and concomitant medications will be reported and documented.

Visit 4 (week 12 ± 7 days) End of Phase 1 During this visit, parents will return the used IP. A clinical and behavioral evaluation will be held via questionnaires (ABC-C, CGI-1, CSHQ and SP-2) and the investigator, vital signs and weight will be measured.

The patient's compliance diary will be reviewed and returned to the parents for further documentation and adverse events and concomitant medications will be reported and documented.

The patient will participate in a 10-minute eye tracking test. Immediately after this visit, a four-week washout period will be initiated and no investigational product will be administered.

Visit 5 (week 16 ± 10) Crossover and Initiation of Phase 2 During this visit, the IP will be crossed over, and those who were first randomized to receive placebo will now receive the product and vice versa.

A clinical and behavioral evaluation will be held by the investigator and will also include the following questionnaires (ABC-C, CGI-1, CSHQ and SP-2), urine sample will be taken for the presence of cannabis and the patient will participate in a 10-minute eye tracking test. In addition, the patient compliance diary will be reviewed and returned to the parents for further documentation and adverse events and concomitant medications will be reported and documented.

A detailed guidance and instructions on the use of the IP at home will be given by a member of the trial team. The first dose administration will be the morning after the visit.

Visit 6 (week 22 ± 5) Mid-Phase 2 During this visit, a clinical and behavioral evaluation will be held via questionnaires (ABC-C, CGI-1) and the investigator. The patient compliance diary will be reviewed and returned to the parents for further documentation. Adverse events and concomitant medications will be reported and documented.

Visit 7 (week 28 ± 7) End of Phase 2 During this visit, parents will return the used IP. A clinical and behavioral evaluation will be held via questionnaires (ABC-C, CGI-1, CSHQ and SP-2) and the investigator. Vital signs and weight will be measured, the patient compliance diary will be returned and adverse events and concomitant medications will be reported and documented.

The patient will participate in a 10-minute eye tracking test. Visit 8 (week 32 ± 14) End of Trial During this visit, a clinical and behavioral evaluation will be held via questionnaires (ABC-C, CGI-1) and the investigator. Vital signs and weight and height will be measured and a urine sample will be taken for the presence of cannabis. Adverse events and concomitant medications will be reported and documented.

EEG Sub-study Parents will receive an explanation regarding the option to participate in an overnight EEG exams performed in the sleep laboratory at SUMC. This test is not mandatory for participation in the trial but will help researches assess the influence cannabis has on brain activity during sleep. Participating children and parents will be invited to three overnight EEG exams throughout the trial: right after enrollment and before initiating the trial (baseline), again right after the end of phase one (week 12-16), and a third and final exam right after the end of phase two (week 28-32).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Children ages two to eight years old with a documented diagnosis of ASD.
* Children with a previous report of behavioral issues characterized by aggression, anxiety, restlessness, sleep disturbances and/or self-harm, all as a part of the ASD, as documented in previous clinical estimation and examination.
* Hebrew speaking and reading.

Exclusion Criteria:

* Children that are treated with cannabis, anti-psychotic drugs or stimulants.
* Children with a comorbidity of heart, liver, kidney or hematologic disease.
* Children that are treated with one of the following drugs: Astemizole, Cisapride, Pimozide or Terfenadine.
* Children that suffer from epilepsy
* Children which themselves or a first-degree family member suffer from psychosis and/or another mental illness.
* Children in any condition in which the investigator is of the opinion that participating in the study is not the best option for them.
* Children who underwent surgery during the 30 days prior to the trial.
* Children that are participating in another trial which includes any intervention.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
change in symptoms of Autism spectrum disorder | 32 weeks
  Superiority in reducing symptoms of Autism spectrum disorder as described and quantified via parent questionnaires and clinical assessment held by a specialized physician, in five main categories - sensory behavior, social relating, body and object use, language and communication skills, and social and adaptive skills. Clinical estimation will be held via the Aberrant Behavior Checklist-Community (ABC-C) questionnaire. Clinical estimation will be performed at the beginning and the end of each phase. Comparison will be held between clinical estimation results after treatment with MCG versus after treatment with placebo for both arms.

SECONDARY OUTCOMES:
change in score of The Clinical Global Impressions-Improvement (CGI-I) | 32 weeks
  Superiority in reducing symptoms of Autism spectrum disorder as described and quantified via parent questionnaire - The Clinical Global Impressions-Improvement (CGI-I). Clinical estimation will be performed at the beginning and the end of each phase. Comparison will be held between clinical estimation results after treatment with MCG versus after treatment with placebo for both arms.
change in score of Sensory Profile II (SP-2) | 32 weeks
  assessed by the Sensory Profile II (SP-2) questionnaire. Parents will answer the questionnaire at the beginning and the end of each trial phase and a comparison will be held within each arm according to baseline and between both arms.
Changes in eye movements | 32 weeks
  tracking as participants observe movies with social information. An eye tracking (ET) experiment will be performed at the beginning and end of each phase to examine changes in the way the children observe movies with social information (e.g. children playing). A comparison will be held within each arm according to baseline and between both arms.
Changes in the sleep architecture (optional) | 32 weeks
  Parents will receive an explanation regarding the option to participate in an overnight EEG exams performed in the sleep laboratory at SUMC. This test is not mandatory for participation in the trial but will help researches assess the influence cannabis has on brain activity during sleep. Participating children and parents will be invited to three overnight EEG exams throughout the trial: right after enrollment and before initiating the trial (baseline), again right SCRC17039 Version 1.1, March 2018 Page 34 of 51 CONFIDENTIAL This material is the property of TO Pharma LLC. The information is confidential and is to be used only in connection with matters authorized by the sponsor and no part of it is to be without prior written permission from TO Pharma LLC.
  after the end of phase one (week 12-16), and a third and final exam right after the end of phase two (week 28-32).

CONTACTS AND LOCATIONS:
Overall Officials: Lihi Bar-LEv, Study Director — Clinical team manager
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No